CLINICAL TRIAL: NCT03415100
Title: Pilot Study of NKG2D-Ligand Targeted CAR-NK Cells in Patients With Metastatic Solid Tumours
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRC-NK-01
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Solid Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-NK cells targeting NKG2D ligands (Experimental)
  Interventions: Biological: CAR-NK cells targeting NKG2D ligands

INTERVENTIONS:
Biological: CAR-NK cells targeting NKG2D ligands — The infusion of CAR-NK cells will be performed in the Third Affiliated Hospital of Guangzhou Medical University. Following infusion of CAR-NK cells, interleukin-2 (IL-2) will be injected subcutaneously into some patients to support the in vivo survival of CAR-NK cells. The subject will be observed for any side effects during this time and all the adverse events will be recorded.

SUMMARY:
This is a single-centre, single arm, open-label pilot study to evaluate the safety and feasibility of CAR-NK cell treatment in subjects with metastatic solid tumours. Autologous or allogeneic NK cells are transfected by mRNA electroporation to prepare investigational CAR-NK cells with transiently enhanced specificity and activity against NKG2D-ligand expressing cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form must be obtained prior to any research procedure.
2. Histologically or cytologically confirmed diagnosis of metastatic solid tumours
3. ECOG performance status of 0-3;
4. Adequate organ function defined as: ANC≥1.0×10^9/L, PLT≥75×10^9/L, ALB≥25g/L, TBIL≤1.5×ULN, AST≤2.5×ULN, ALT≤2.5×ULN, ALP≤2.5×ULN, Cr≤1.5×ULN;
5. The patient's own PBMCs or PBMCs from a biological parent or child who is willing to donate blood will be used to prepare CAR-NK cells. The parent or child should be ≥18 and ≤60 years old, and he or she is able to sign the informed consent for blood donation by himself/herself;
6. Patients who won't benefit from surgery, or refuse surgical treatment; patients who won't benefit from chemotherapy, can't tolerate chemotherapy or refuse chemotherapy.
7. Patients volunteer to participate in this study and sign the informed consent form for subjects;
8. Blood donors sign the informed consent form for blood donors.
9. Blood donors have negative test results for HIV, HBV and HCV;
10. If a subject or blood donor is a female of childbearing potential, she must have a negative urine pregnancy test result.

Exclusion Criteria:

1. Patients who are suffering from uncontrollable or active infectious diseases of the hematological system, cardiovascular system, respiratory system, digestive system, urinary system, or the endocrine system;
2. Patients with immunologic deficiency or autoimmune diseases;
3. Patients with severe hypersensitivity reactions;
4. Patients received other forms of cellular therapies within the last 3 months;
5. Patients received systemic steroids within the last 3 months;
6. Patients who are breastfeeding or pregnant;
7. Patients with brain metastases;
8. Patients who have received an organ transplant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | from day 0 - month 4

SECONDARY OUTCOMES:
Anti-tumour response due to CAR-NK cell infusions | 100 days after CAR-NK cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Xuehu Xu, MD, Principal Investigator — The Third Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Ng YY, Du Z, Zhang X, Chng WJ, Wang S. CXCR4 and anti-BCMA CAR co-modified natural killer cells suppress multiple myeloma progression in a xenograft mouse model. Cancer Gene Ther. 2022 May;29(5):475-483. doi: 10.1038/s41417-021-00365-x. Epub 2021 Sep 1. PMID 34471234